CLINICAL TRIAL: NCT04234321
Title: A Multicenter, Prospective Clinical Study of Kangfuxin and Basic Fibroblast Growth Factor in Promoting the Healing of Donor Site
Brief Title: Clinical Study of Kangfuxin and Basic Fibroblast Growth Factor in Promoting the Healing of Donor Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); Jiangyin Hospital Affiliated to Southeast University School of Medicine (Unknown); Nantong University (Other); The 59th Central Hospital of the Chinese people's Liberation Army (Unknown); Taizhou Hospital (Other); Zhejiang Quhua Hospital (Other); Lishui Country People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR201900069
Record Dates: First submitted 2020-01-04; First posted 2020-01-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-01

CONDITIONS: Fibroblast Growth Factors; Wound Healing
Keywords: basic fibroblast growth factor,Kangfuxin,Wound Healing
MeSH Terms: interventions — Fibroblast Growth Factor 2; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- basic fibroblast growth factor (Experimental): Basic fibroblast growth factor,100ml/ bottle, (35000IU / 8ml) / 100cm2 / time,three times a day.
  Interventions: Drug: basic fibroblast growth factor
- Kangfuxin Liquid (Experimental): Kangfuxin Liquid,20ml / 100cm2 / time,three times a day.
  Interventions: Drug: Kangfuxin Liquid
- 0.9% Normal saline (Placebo Comparator): 0.9% Normal saline,20ml / 100cm2 / time,three times a day.
  Interventions: Drug: 0.9% Normal saline

INTERVENTIONS:
Drug: basic fibroblast growth factor — Basic fibroblast growth factor,100ml/ bottle, (35000IU / 8ml) / 100cm2 / time,three times a day.
  Arms: basic fibroblast growth factor
Drug: Kangfuxin Liquid — Kangfuxin Liquid,20ml / 100cm2 / time,three times a day.
  Arms: Kangfuxin Liquid
Drug: 0.9% Normal saline — 0.9% Normal saline,20ml / 100cm2 / time,three times a day.
  Arms: 0.9% Normal saline

SUMMARY:
The main objective of this study is to observe whether basic fibroblast growth factor and Kangfuxin Liquid can promote the wound healing in the donor area and further evaluate the healing quality.

ELIGIBILITY:
Inclusion Criteria:

* Male / female patients aged 20-50;
* Burn area ≤ 30% TBSA;
* Patients who need auto skin grafting due to burns or skin defects due to trauma;
* The donor area is 100cm2, and the thickness of skin is 0.25mm (Split thickness skin donor site group)/0.40mm (Medium thickness skin donor site group). The donor site is the body part with similar skin color and sufficient skin area (except scalp);
* Not involved in clinical trials of other drugs;
* Subjects who have agreed to participate in the clinical study and signed the informed consent.

Exclusion Criteria:

* Subjects who were previously allergic to similar products or related components of test products;
* Subjects with other systemic or local skin diseases that may affect wound evaluation;
* Subjects with significant organ dysfunction / failure or other serious diseases, including clinical related cardiovascular disease or myocardial infarction within 12 months before enrollment; malignant tumor; serious neurological or psychiatric history; serious infection; active disseminated intravascular coagulation;
* Subjects with moderate malnutrition (BMI < 17kg / m2) and severe anemia (HB < 60g / L);
* Subjects proposed to use immunosuppressant, steroid hormone, epidermal growth factor and other drugs that may affect the wound healing of the donor skin within 3 months before admission or during the study period;
* Participated in clinical trials of any other drugs or medical devices within 3 months;
* History of major diseases that may affect general physical condition and other patients who are not considered by the researchers to be eligible for this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate | up to 2 or 3 weeks
  Means (wound area before treatment - wound area after treatment) / wound area before treatment × 100%.
Actual healing time | up to 2 or 3 weeks
  Means time of complete wound healing

SECONDARY OUTCOMES:
Degree of scar formation | up to 3 or 12 weeks
  The degree of scar formation .

CONTACTS AND LOCATIONS:
Overall Officials: huawei shao, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China